CLINICAL TRIAL: NCT00066027
Title: Low-Dose Doxycycline Effects on Osteopenic Bone Loss
Brief Title: Effects of Low-Dose Doxycycline on Oral Bone Loss
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Nebraska (Other)
Collaborators: National Institute of Dental and Craniofacial Research (NIDCR) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 0511-00-FB; R01DE012872 (NIH)
Record Dates: First submitted 2003-08-01; First posted 2003-08-05 (Estimated); Last update posted 2023-09-06 (Actual); Status verified 2023-09

CONDITIONS: Periodontitis
Keywords: periodontitis, metabolic bone diseases, doxycycline
MeSH Terms: conditions — Periodontitis; Bone Diseases, Metabolic | interventions — Doxycycline; Anti-Bacterial Agents; Sugars

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- low-dose doxycycline (Experimental): low-dose doxycycline (20 mg doxycycline hyclate)
  Interventions: Drug: 20 mg doxycycline hyclate
- Placebo (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: 20 mg doxycycline hyclate — Subjects in the LDD group took 20 mg doxycycline hyclate tablets twice daily for two years
  Other Names: antibiotic
  Arms: low-dose doxycycline
Drug: Placebo — Subjects in the placebo group took a placebo look-alike twice daily for two years.
  Other Names: sugar pill
  Arms: Placebo

SUMMARY:
The primary purpose of this clinical trial is to determine whether low-dose doxycycline can reduce alveolar bone density loss in postmenopausal osteopenic women with periodontitis and not on hormone replacement therapy (i.e., estrogen deficient).

DETAILED DESCRIPTION:
The primary purpose of this clinical trial is to determine whether low-dose doxycycline (LDD) can reduce alveolar bone density loss in postmenopausal osteopenic women with periodontitis and not on hormone replacement therapy (i.e., estrogen deficient). The effects of LDD on alveolar bone height loss, progressive periodontal attachment loss, systemic bone mineral density, gingival crevicular fluid biochemical markers of collagen degradation and bone resorption and serum biomarkers of bone formation, bone resorption and inflammation also will be assessed. In addition, another objective is to determine if the microbial effects obtained with LDD over two years are equivalent to a placebo control. This clinical trial involves two clinical sites: the University of Nebraska Medical Center College of Dentistry and Stony Brook University School of Dental Medicine. A total of 128 postmenopausal osteopenic women with periodontitis between the ages of 45 and 70 at the time of telephone screening will be randomized to LDD or placebo groups and subjects will be followed for two years.

ELIGIBILITY:
Inclusion Criteria:

* Subjects will be female, postmenopausal and not receiving estrogen replacement therapy.
* Subjects will be 45-70 years old at the time of telephone screening.
* Subjects will have osteopenia (T-score of -1.0 to -2.5) of the lumbar spine or femoral neck as determined by dual-energy absorptiometry (DEXA) scans.
* Subjects will have a history of generalized moderate-advanced periodontitis and will be undergoing periodontal maintenance.
* Subjects will be in good general health and willing to sign the IRB-approved consent form.

Exclusion Criteria:

* Subjects will not have an allergy or hypersensitivity to tetracyclines.
* Subjects will not have diseases or take medications that affect the inflammatory or immune responses (e.g., chronic use of non-steroidal anti-inflammatory drugs) or bone remodeling (e.g., drugs such as prescription estrogens, bisphosphonates, calcitonin or steroids).
* Subjects will not have any medical condition requiring antibiotic premedication (e.g., prosthetic heart valves, prosthetic joints, and mitral valve prolapse with regurgitation) for routine dental therapy.
* Subjects cannot have diabetes mellitus.
* Subjects cannot have had active periodontal therapy (quadrant scaling and root planing or periodontal surgery) within the past year.
* Subjects cannot have osteoporosis (T-score greater than -2.5) of the lumbar spine or femoral neck.

Ages: 45 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 128 (Actual)
Dates: Start 2002-06-01 (Actual); Primary Completion 2005-10-01 (Actual); Study Completion 2005-10-01 (Actual)

PRIMARY OUTCOMES:
Alveolar Bone Density | Baseline, one-year and two-year visits
  Alveolar bone density changes assessed by radiographic absorptiometry and computer-assisted densitometric image analysis.

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey B Payne, DDS, Principal Investigator — UNMC College of Dentistry
Locations (2):
- United States (2):
  - University of Nebraska Medical Center, College of Dentistry, Lincoln, Nebraska
  - Department of Oral Biology and Pathology, Stony Brook, New York

REFERENCES:
- [Background] Stoner JA, Payne JB. Interpretation of treatment effects in periodontal research: a note on the number needed to treat. J Can Dent Assoc. 2008 Jun;74(5):435-7. No abstract available. PMID 18538066
- [Result] Salminen A, Pussinen PJ, Payne JB, Stoner JA, Jauhiainen M, Golub LM, Lee HM, Thompson DM, Sorsa T. Subantimicrobial-dose doxycycline treatment increases serum cholesterol efflux capacity from macrophages. Inflamm Res. 2013 Jul;62(7):711-20. doi: 10.1007/s00011-013-0626-z. Epub 2013 May 7. PMID 23649042
- [Result] Payne JB, Nummikoski PV, Thompson DM, Golub LM, Stoner JA. The association between clinical and radiographic periodontitis measurements during periodontal maintenance. J Periodontol. 2013 Oct;84(10):1382-90. doi: 10.1902/jop.2012.120484. Epub 2012 Dec 3. PMID 23205917
- [Result] Gu Y, Walker C, Ryan ME, Payne JB, Golub LM. Non-antibacterial tetracycline formulations: clinical applications in dentistry and medicine. J Oral Microbiol. 2012;4. doi: 10.3402/jom.v4i0.19227. Epub 2012 Oct 12. PMID 23071896
- [Result] Payne JB, Golub LM, Stoner JA, Lee HM, Reinhardt RA, Sorsa T, Slepian MJ. The effect of subantimicrobial-dose-doxycycline periodontal therapy on serum biomarkers of systemic inflammation: a randomized, double-masked, placebo-controlled clinical trial. J Am Dent Assoc. 2011 Mar;142(3):262-73. doi: 10.14219/jada.archive.2011.0165. PMID 21357860
- [Result] Payne JB, Golub LM. Using tetracyclines to treat osteoporotic/osteopenic bone loss: from the basic science laboratory to the clinic. Pharmacol Res. 2011 Feb;63(2):121-9. doi: 10.1016/j.phrs.2010.10.006. Epub 2010 Oct 16. PMID 20937388
- [Result] Golub LM, Lee HM, Stoner JA, Reinhardt RA, Sorsa T, Goren AD, Payne JB. Doxycycline effects on serum bone biomarkers in post-menopausal women. J Dent Res. 2010 Jun;89(6):644-9. doi: 10.1177/0022034510363367. Epub 2010 Mar 26. PMID 20348487
- [Result] Reinhardt RA, Stoner JA, Golub LM, Lee HM, Nummikoski PV, Sorsa T, Payne JB. Association of gingival crevicular fluid biomarkers during periodontal maintenance with subsequent progressive periodontitis. J Periodontol. 2010 Feb;81(2):251-9. doi: 10.1902/jop.2009.090374. PMID 20151804
- [Result] Golub LM, Lee HM, Stoner JA, Sorsa T, Reinhardt RA, Wolff MS, Ryan ME, Nummikoski PV, Payne JB. Subantimicrobial-dose doxycycline modulates gingival crevicular fluid biomarkers of periodontitis in postmenopausal osteopenic women. J Periodontol. 2008 Aug;79(8):1409-18. doi: 10.1902/jop.2008.070623. PMID 18672990
- [Result] Walker C, Puumala S, Golub LM, Stoner JA, Reinhardt RA, Lee HM, Payne JB. Subantimicrobial dose doxycycline effects on osteopenic bone loss: microbiologic results. J Periodontol. 2007 Aug;78(8):1590-601. doi: 10.1902/jop.2007.070015. PMID 17668979
- [Derived] Payne JB, Stoner JA, Lee HM, Nummikoski PV, Reinhardt RA, Golub LM. Serum bone biomarkers and oral/systemic bone loss in humans. J Dent Res. 2011 Jun;90(6):747-51. doi: 10.1177/0022034511402993. Epub 2011 Mar 21. PMID 21422479
- [Derived] Payne JB, Stoner JA, Nummikoski PV, Reinhardt RA, Goren AD, Wolff MS, Lee HM, Lynch JC, Valente R, Golub LM. Subantimicrobial dose doxycycline effects on alveolar bone loss in post-menopausal women. J Clin Periodontol. 2007 Sep;34(9):776-87. doi: 10.1111/j.1600-051X.2007.01115.x. PMID 17716313
- [Derived] Reinhardt RA, Stoner JA, Golub LM, Wolff MS, Lee HM, Meinberg TA, Lynch JC, Ryan ME, Sorsa T, Payne JB. Efficacy of sub-antimicrobial dose doxycycline in post-menopausal women: clinical outcomes. J Clin Periodontol. 2007 Sep;34(9):768-75. doi: 10.1111/j.1600-051X.2007.01114.x. PMID 17716312